CLINICAL TRIAL: NCT02753725
Title: Effect of Fentanyl Given Approximately Ten Minutes to the End of Surgery on Emergence Delirium in Children Undergoing Adeno-tonsilectomy at Kenyatta National Hospital: A Randomized Placebo Controlled Clinical Trial
Brief Title: Effect of Fentanyl on Emergence Delirium (ED) on Children Undergoing Adeno-tonsilectomy at Kenyatta National Hospital (KNH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nairobi (Other)
Responsible Party: Principal Investigator, Dr. Kirwa Elisha kiprono, Dr., University of Nairobi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UNairobi 1
Record Dates: First submitted 2016-04-11; First posted 2016-04-28 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Fentanyl; Therapeutics; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl group (Active Comparator): Fentanyl given at a dose of one micro gram per kilogram body weight
  Interventions: Drug: Fentanyl
- normal saline group (Placebo Comparator): placebo arm will be given normal saline at a volume equivalent to Fentanyl dose as per body weight.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Fentanyl — The intervention arm will comprise Fentanyl given at a dose of one microgram per kilogramme body weight administered approximately ten minutes to the end of surgery determined by the time when the mouth gag will be removed.
  Other Names: treatment
  Arms: Fentanyl group
Drug: Normal saline — the placebo arm will be given normal saline at a volume equivalent to Fentanyl dose per body weight,administered approximately ten minutes to the end of surgery determined by the time when the mouth gag will be removed
  Other Names: placebo
  Arms: normal saline group

SUMMARY:
This study will be a randomized double blind placebo controlled clinical trial among children undergoing adeno-tonsillectomy in KNH. The intervention arm will comprise Fentanyl given at a dose of 1ug/while the placebo arm will be given normal saline at a volume equivalent to Fentanyl dose, treatment will be administered approximately ten minutes to the end of surgery determined by the time when the mouth gag will be removed. The main outcome will be incidence of ED at the recovery room using Watcha scale and secondary outcomes will be delay in emergence time from anaesthesia and effectiveness of fentanyl in preventing ED.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists classes (ASA) 1 and 2 children.

  * ASA 1 - Normal healthy child scheduled for adeno-tonsilectomy.
  * ASA 2 - Child with mild systemic disease without functional limitations.
* Children aged 1 to 12 years.
* Children undergoing elective adeno-tonsilectomy.
* Those children whose parents/guardians have given a written informed consent.

Exclusion Criteria:

* Children with genetic syndromes.
* Children with psychological/neurological behavioural disorders.
* Children with allergies to Fentanyl.
* Children with psychiatric disorders/ use of psychiatric medications.
* Use of sedative medications one hour prior to surgery.
* Children with developmental delay.
* Children coming in as day case.
* Children with airway problems not related to the surgery-sleep apnoea.
* Children less than 1 year and those above 13 years.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The number of patients who develop emergence delirium in both arms | 30 minutes
  the number of patients who develop emergence delirium within 30 minutes after general anaesthesia will be assessed using Watcha scale indicated in the study questionnaire,
the local incidence of emergence delirium. | 30 minutes
  local incidence of emergence delirium will be determined by the percentage of those who develop emergence delirium in the placebo group within 30 minutes after general anesthesia as assessed by Watcha scale.

SECONDARY OUTCOMES:
the percentage of patients developing emergence delirium in fentanyl group with 30 minutes after general anaesthesia. | 30 minutes
  the percentage of patients developing emergence delirium in both groups will be compared to determine if fentanyl prevents emergence delirium.
duration of emergence time from general anaesthesia in minutes | 30 minutes
  the time taken to emerge from both arms will be compared to determine if fentanyl delays emergence time from general anaesthesia.

IPD SHARING:
Plan to Share IPD: Yes
conferences, report writing